CLINICAL TRIAL: NCT01574183
Title: Vilazodone Treatment for Marijuana Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Aimee McRae-Clark, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16488; R21DA034089 (NIH)
Record Dates: First submitted 2012-04-05; First posted 2012-04-10 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-07

CONDITIONS: Marijuana Dependence
Keywords: Marijuana; Vilazodone; Contingency management; Motivational enhancement therapy
MeSH Terms: conditions — Marijuana Abuse | interventions — Vilazodone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vilazodone (Experimental): Flexible dose up to 40 mg capsule daily
  Interventions: Drug: Vilazodone
- Placebo (Placebo Comparator): Flexible dose up to 40 mg capsule daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vilazodone — up to 40 mg capsule daily
  Other Names: Viibryd
  Arms: Vilazodone
Drug: Placebo — up to 40 mg capsule daily
  Arms: Placebo

SUMMARY:
Marijuana is the most commonly used illicit drug, yet few clinical trials have evaluated pharmacotherapy treatments for marijuana dependence. This study will evaluate the efficacy of vilazodone for reducing marijuana use in marijuana-dependent adults. A contingency management intervention (CM)and motivational enhancement therapy (MET)will be incorporated to encourage study engagement and retention, and genomic DNA will be extracted to characterize subjects according to polymorphisms of genes potentially relevant to the activity of vilazodone. It is hypothesized that vilazodone combined with MET and CM will reduce the percent of marijuana-positive urine drug screen results in marijuana-dependent individuals as compared to a placebo treatment combined with MET and CM.

DETAILED DESCRIPTION:
The purpose of this study is to determine if the medication vilazodone is effective in helping frequent marijuana smokers cut down or stop using marijuana. Vilazodone is FDA approved for the treatment of depression- in this study, vilazodone's effect on marijuana dependence is being investigated.

Participation in the study takes 10 visits over a period of approximately two to three months. The first visit is a screening visit to determine if participants are eligible to participate. After the initial assessment visit, the weekly visits take about 30 minutes, with the exception of three therapy sessions which take approximately 60-90 minutes. The three therapy sessions will focus on participant's marijuana use and reasons they may have for stopping or cutting down on use. After completing an initial therapy session, participants will be randomly selected to receive the study medication, either vilazodone or placebo (a capsule that does not contain any active medication). Participants will have weekly study visits with a clinician. At each study visit, they will be asked to fill out forms and answer specific questions concerning their substance use, anxiety symptoms, and feelings in general. They will be providing urine samples to check for illegal drugs of abuse including marijuana and other drugs. They will also have blood samples drawn during to determine if you are taking the medication as directed.

ELIGIBILITY:
Inclusion Criteria:

* Must meet DSM-IV criteria for marijuana dependence
* Must be between the ages of 18 and 65 years old
* If female and of childbearing potential, must agree to use acceptable method of birth control for duration of the trial.
* Cannabis-positive urine drug screen at screening
* Must consent to random assignment
* Must be able to read and provide informed consent

Exclusion Criteria:

* Women who are pregnant, nursing, or plan to become pregnant during course of study
* Must not have a history of or current psychotic disorder, bipolar disorder, or eating disorder
* Must not pose a current suicidal or homicidal risk
* Must not have evidence or history of serious medical disease
* Must not require concomitant therapy with psychotropic medication or CYP3A4 inhibitors
* Must not be currently dependent on other substances, with the exception of nicotine;
* Patients who, in the investigator's opinion, would be unable to comply with study procedures or assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-08; Primary Completion 2015-08 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee L McRae-Clark, PharmD, BCPP, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited between August, 2012 and August, 2014 primarily through media and internet advertisements.
Groups:
- Vilazodone: Flexible dose up to 40 mg capsule daily
  Vilazodone: 40 mg capsule daily
- Placebo: Flexible dose up to 40 mg capsule daily
  Placebo: 40 mg capsule daily
Period: Overall Study
Arm/Group | Vilazodone | Placebo
Started | 41 | 35
Completed | 14 | 17
Not Completed | 27 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vilazodone | Placebo | Total
Number analyzed (Participants) | 41 | 35 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 35 | 76
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 30 | 30 | 60
Region of Enrollment [Number; unit: participants]
  United States | 41 | 35 | 76

OUTCOME MEASURES:

1. Primary Outcome: Percent Marijuana-negative Urine Drug Screens (UDS)
Description: Participants submitted a urine sample weekly. Percentage of marijuana negative urine samples were calculated per group.
Time Frame: 8 weeks
Measure: Number; unit: percentage of UDS
Units Other Than Participants: Urine samples
Arm/Group | Vilazodone | Placebo
Number analyzed (Participants) | 41 | 35
Number analyzed (Urine samples) | 328 | 280
percentage of UDS | 5.5 | 3.6

2. Secondary Outcome: Weekly Cannabis Use Sessions
Description: Self-report of weekly cannabis use sessions was measured using the Time Line Followback, a calendar-based instrument designed to assess substance consumption.
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: weekly cannabis sessions
Arm/Group | Vilazodone | Placebo
Number analyzed (Participants) | 41 | 35
weekly cannabis sessions | 10 [8.1 to 11.8] | 9.9 [8.2 to 11.7]

3. Secondary Outcome: Marijuana Craving and Withdrawal
Description: The Marijuana Craving Questionnaire (MCQ) is intended to measure marijuana craving in adults. It measures symptoms on four subscales: expectancy, purposefulness, emotionality, and compulsivity. The scale rates individual items from 1 (least craving) - 7 (most craving) with a composite scoring range of 12-84 and possible subscale scoring range of 3-21. It was administered weekly to all participants. Reported here is the mean MCQ purposefulness subscale score across 8 weeks.
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Vilazodone | Placebo
Number analyzed (Participants) | 41 | 35
units on a scale | 8.9 [7.5 to 10.3] | 11.3 [9.9 to 12.7]

ADVERSE EVENTS:
Groups:
- Vilazodone: Flexible dose Vilazodone: up to 40 mg capsule daily
- Placebo: Flexible dose Placebo: up to 40 mg capsule daily
Arm/Group | Vilazodone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/35
Other Adverse Events (participants affected / at risk) | 25/41 | 28/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vilazodone (N=41) | Placebo (N=35)
Allergies (General disorders) | 1 (1) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 5 (10) | 3 (3)
Dizzy/lightheaded (Nervous system disorders) | 4 (5) | 2 (2)
Dream disturbance (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 8 (12) | 4 (10)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 5 (7) | 6 (6)
Nausea (Gastrointestinal disorders) | 13 (17) | 5 (8)
Other GI (Gastrointestinal disorders) | 3 (3) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Vomiting (Gastrointestinal disorders) | 5 (8) | 0 (0)
Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (9)
Insomnia (Nervous system disorders) | 4 (5) | 5 (5)
Other (General disorders) | 10 (17) | 10 (13)

LIMITATIONS AND CAVEATS:
Limitations included small sample size, significant attrition, and difficulty with UCT (urine cannabinoid test) interpretation due to long excretion half-life of cannabis in urine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No